CLINICAL TRIAL: NCT05240066
Title: Birth Control to Improve Birth Spacing: a Prospective Longitudinal Cohort Study
Brief Title: Birth Control to Improve Birth Spacing
Acronym: BIBS
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Boston Medical Center (Other); Harvard Medical School (HMS and HSDM) (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Elizabeth Janiak, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 2021P000762; R21HD103977 (NIH)
Record Dates: First submitted 2022-01-20; First posted 2022-02-15 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Contraception; Contraception Behavior; Knowledge, Attitudes, Practice; Birth Spacing
Keywords: birth spacing; behavior; environmental barriers; pospartum; contraception
MeSH Terms: conditions — Contraception Behavior; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the drivers of postpartum contraceptive use with a prospective cohort. The study will clarify the role of contraceptive knowledge, attitudes, norms, and self-efficacy in driving intention to initiate contraception postpartum and describe the impact of environmental barriers on enacting intended postpartum contraception initiation.

DETAILED DESCRIPTION:
This study will be a sequential mixed-methods design with a prospective cohort to identify and explore barriers to contraceptive initiation both immediately after birth and prior to hospital discharge, as well as throughout the fourth trimester. It will include a baseline patient survey, electronic medical record data pull, follow up survey, and qualitative interviews.

The investigators will enroll 1400 patients into the prospective cohort, selecting individuals enrolled at prenatal care visits at two sites. The baseline survey will be self-administered. The investigators will then contact participants for a follow-up survey at 12 weeks postpartum. Surveys will be self-administered through a link received by text message or email. Additional analyses will draw on retrospectively collected medical record data.

The investigators will invite a subset of 25-30 study subjects to participate in qualitative interviews.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Pregnant
* Attending prenatal care visits at one of the two study sites

Exclusion Criteria:

* Under the age of 18
* Cannot complete a survey in English or Spanish
* Do not have physical or cognitive ability to complete a survey on a tablet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will enroll 1,400 patients into the prospective cohort, selecting individuals enrolled at prenatal care visits at Boston Medical Center and Brigham and Women's Hospital main campus. All subjects enrolled in the baseline survey who deliver at enrollment sites will be included in electronic medical records and contacted for a follow-up survey at 12 weeks postpartum.
  Additionally, the investigators will invite a subset of the study subjects (25-30 patients) who report significant barriers to contraceptive uptake in the 12-week postpartum follow up survey to participate in qualitative interviews.
Sampling Method: Non-Probability Sample
Enrollment: 1341 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Desired birth spacing | Baseline
  self-reported desire to space births
Contraceptive attitudes and norms | Baseline
  measured via validated psychometric scales; Examining Contraceptive Use and Unmet Need Study, 12-58 range, higher score indicates more knowledge, citation: Callegari, Lisa S., MD, MPH, Zhao, Xinhua, PhD, Schwarz, Eleanor Bimla, MD, MS, Rosenfeld, Elian, PhD, Mor, Maria K., PhD, & Borrero, Sonya, MD, MS. (2017). Racial/ethnic differences in contraceptive preferences, beliefs, and self-efficacy among women veterans. American Journal of Obstetrics and Gynecology, 216(5), 504.e1-504.e10.
  DOI: 10.1016/j.ajog.2016.12.178
contraceptive self-efficacy | Baseline
  measured via validated psychometric scales; Examining Contraceptive Use and Unmet Need Study, 12-58 range, higher score indicates more knowledge, citation: Callegari, Lisa S., MD, MPH, Zhao, Xinhua, PhD, Schwarz, Eleanor Bimla, MD, MS, Rosenfeld, Elian, PhD, Mor, Maria K., PhD, & Borrero, Sonya, MD, MS. (2017). Racial/ethnic differences in contraceptive preferences, beliefs, and self-efficacy among women veterans. American Journal of Obstetrics and Gynecology, 216(5), 504.e1-504.e10.
  DOI: 10.1016/j.ajog.2016.12.178
Contraceptive knowledge | Baseline
  measured via the Contraceptive Knowledge Assessment (Haynes et al 2017), 0-25 score range, higher scores reflect greater knowledge. Haynes MC, Ryan N, Saleh M, Winkel AF, Ades V. Contraceptive Knowledge Assessment: validity and reliability of a novel contraceptive research tool. Contraception. 2017 Feb;95(2):190-197. doi: 10.1016/j.contraception.2016.09.002. Epub 2016 Sep 9.
Intention to initiate contraception postpartum | Baseline
  self-reported desire to use contraception within 12 weeks of birth
Planned postpartum contraceptive method | Baseline
  self-report of selected method
Contraceptive use | 12-week follow up
  Participants will be asked if they have used a contraceptive method since giving birth.
Environmental barriers to contraceptive use | 12-week follow up
  Participants will rate the difficulty in accessing their desired contraceptive method after giving birth and respond to the reasons why it is - or is not - easy to access.

SECONDARY OUTCOMES:
Intimate partner violence | 12-week follow up
  measured via validated psychometric scales; Abuse Assessment Screen, 5 items, citation: Soeken, K. L., McFarlane, J., Parker, B., & Lominack, M. C. (1998). The Abuse Assessment Screen: A clinical instrument to measure frequency, severity, and perpetrator of abuse against women. In J. C. Campbell (Ed.), Sage series on violence against women. Empowering survivors of abuse: Health care for battered women and their children (pp. 195-203). Thousand Oaks, CA, US: Sage Publications, Inc.

OTHER OUTCOMES:
Immediate and delayed postpartum method uptake | 72 hours postpartum, 12 weeks postpartum
  contraceptive method prescribed, inserted, injected, or otherwise provided

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available.